CLINICAL TRIAL: NCT06906094
Title: Prevention of Post mEniscectomy Osteoarthritis: From New Animal Model to Patient pRofiLing (PEARL)
Brief Title: Prevention of Post mEniscectomy Osteoarthritis: From New Animal Model to Patient pRofiLing
Acronym: PEARL
Status: Enrolling by invitation | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other); Azienda Ospedaliero Universitaria di Sassari (Other)
Responsible Party: Sponsor
Other Study IDs: Protocol ID: 2801 Study N:3421
Record Dates: First submitted 2025-03-18; First posted 2025-04-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Meniscopathy
Keywords: meniscectomy; surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Before surgery, peripheral blood samples from each patient enrolled in the observational study will be collected. Total blood count will be registered and included in the set of the patients' data. Total RNA will be purified from the blood samples and integrity of each RNA sample will be evaluated to esclude possible degradation during the procedure. Total RNA will be preamplified to perform the qRT-PCR-based analysis sifting a well-described set of 754 miRNAs panel known for their involvement in several joint and blood cell types' homeostasis and activation. The most abundantly expressed and relevant miRNAs will be identified in the whole set of samples and included in the set of the patients' data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Selective meniscectomy — involves the partial removal of the damaged meniscus.

SUMMARY:
Data collection from patients included in the observational clinical study will be achieved by the following activities:

A total of 100 patients with degenerative meniscal tears will be enrolled in the observational study and treated according to the current standard of care which consists in an arthroscopic partial meniscectomy in all the three clinical operative Unit involved in the project.

Demographic, anamnestic and clinical data (age, gender, BMI, habits, co-morbidities, pharmacological treatments) of the patients included in the observational clinical study will be collected.

Clinical routine assessments will be performed before surgery to assess the overall condition of the joint. A morphological profiling based on the MRI will be performed on patients prior or after the surgery since no change in knee morphology is expected to occur. Clinical routine assessments will be performed also after treatment to check for possible joint changes after the surgery.

Before surgery, peripheral blood samples from each patient enrolled in the observational study will be collected. Total blood count will be registered and included in the set of the patients' data. Total RNA will be purified from the blood samples and integrity of each RNA sample will be evaluated to exclude possible degradation during the procedure.Total RNA will be preamplified to perform the qRT-PCR-based analysis sifting a well-described set of 754 miRNAs panel known for their involvement in several joint and blood cell types' homeostasis and activation. The most abundantly expressed and relevant miRNAs will be identified in the whole set of samples and included in the set of the patients' data. Combination and interpretation of the clinical, morphological, imaging and biomarker -omics data will follow in order to identify the patient characteristics that are more associated to the development of post-meniscectomy OA, following these steps: A patient registry (PEARL registry) containing all the anamnestic, clinical, radiological and morphological data, as well as the blood count and the most relevant and abundant miRNAs obtained through the transcriptomic analyses carried out during the study, will be generated.

Patients will be clinically and radiologically monitored at short- and long-term to evaluate the possible onset of OA post-meniscectomy. Any possible relevant clinical data and adverse events encountered during the patient's clinical path will be tracked.

Patients will be assigned to categories based on the PEARL registry data and their clinical outcome post- meniscectomy. This will help identifying possible risk factors and pre-treatment markers associated to the susceptibility of patients to develop post-meniscectomy OA.

An algorithm that will use the information gathered in the previous steps will be developed. This tool will allow to identify patients more likely to suffer from post-meniscectomy OA and therefore to help in the therapeutic choice. The constant updating of the register over time beyond the project duration will allow to obtain increasingly reliable and consolidated information to further strength the predictivity of the algorithm for choosing the best treatment based on the patients' characteristics.

DETAILED DESCRIPTION:
Patient demographic, anamnestic, clinical, radiological and morphological data will be collected and reported in the database PEARL, assigning an individual ID to each patient. The most relevant and abundant miRNAs obtained through the transcriptomic analyses will be included too. Information about age, gender, body mass index, type of meniscal lesion, type of injury (if any), time of symptoms onset, general knee condition, previous surgical and/or pharmacological treatments, co-morbidities will be included too. Subjective knee evaluations of patients will be collected by using internationally accepted PROMs (Patient Reported Outcome Measures) among which IKDC (International Knee Documentation Committee) Objective Score, KOOS (Knee Injury and Osteoarthritis Outcome Score), VAS (Visual Analogue Score) Pain and EQ-5D-5L. All these data will be collected during the pre-surgical visit and on follow up. Two MRIs are planned for the study, during screening visit and at 6 months follow-up visit; at least one of the two MRIs will be performed with a 3D protocol to assess the bone component. Therefore,radiological and morphological data will include standard x-ray and MRI protocol implemented by metadata of 3D MRI protocol (near-isotropic 0.83mm T2 SPACE and near-isotropic 0.63mm proton density SPACE) when needed. Accurate 3D models of femur bone and cartilage, tibia bone and cartilage and menisci will be reconstructed from (near-)isotropic high-resolution 3D MRI scans. For morphology analysis, a 3D DESS MRI sequence will be complemented with modern clinical sequences for diagnostic purposes. Using the reconstructed 3D models, advanced landmark-based and statistical shape analyses will be performed. The extracted shape features from these analyses will then serve as input for conventional statistical algorithms or state-of-the-art machine learning techniques. Finally, the addition of standing full-leg radiographs gives more insights in the biomechanics of the complete lower-limb from hip to toe. Alignment of the femur with respect to the tibia will be evaluated in both coronal and sagittal plane. These alignment variables will then be used as input for conventional statistics and machine learning algorithms both separately and combined with the knee-specific shape features (cf. previous paragraph).

Data related to the high-throughput transcriptomic analyses will include the most expressed blood miRNAs for each patients. Data will be generated on the Applied Biosystems' QuantStudio' 12K Flex RealTime PCR System using Expression Suite Software. Quantitation will be assessed by the 'relative threshold' method (Crt method) that sets a threshold for each amplification individually that is based on the shape of the amplification curve. Data normalization will be performed with RefFinder tool that evaluates and screens stable candidates from extensive experimental datasets.

After publication, the raw data related to in vitro analyses as well as pre-clinical and clinical anonimazed data will be made available through an open access database.

The timing of analysis data of the study will be as follows:

1. Enrollment and treatment of 100 patients with symptomatic degenerative meniscal lesions undergoing partial arthroscopic meniscectomy: 0-12 months.
2. Transcriptomic analysis will be conducted on blood samples collected at the time of surgery from the patients enrolled in the observational clinical study. The final data will be available within six months after the last enrollment.
3. Follow up evaluation: all the patients will be evaluated at 6 and 12 months. The PEARL registry will permit to eventually clinically and radiologically evaluate the patients also beyond the project duration to monitor the possible onset of post-meniscectomy OA also beyond the one year time limit. Their evaluation after the end of the project will strengthen the findings of the study with longer-term evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form;
2. Male or female patients ≥18 years of age at time of screening;
3. Patients physically and mentally able to comply with all aspects of the study, including the requirements for follow-up visits;
4. Patients suffering from symptomatic medial and/or lateral degenerative meniscal lesion identified at MRI with a surgical indication of arthroscopic partial meniscectomy;
5. In case of bilateral degenerative meniscus, patients with no or mild pain in the contralateral knee, defined as a score < 2 on a 0-10 numerical rating scale (NRS);
6. Patients who, before the last 3 months, have undergone and failed at least one prior conservative OA treatment (NSAIDs, physiotherapy, hydrokinesitherapy);
7. Body mass index (BMI) ≤ 40 kg/m2

Exclusion Criteria:

1. Presence of clinically observed active infection in the index knee joint or skin disease/breakdown or infection in the area of the planned injection site of the index knee
2. Patients who experienced traumatic injury at the index knee within 6 months prior to the procedure;
3. Patients with a history of invasive malignancies (except non- melanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for 5 years;
4. Patients with known systemic disorders or any systemic inflammatory condition such as rheumatoid arthritis;
5. Patients with known metabolic bone diseases such as those affecting calcium metabolism;
6. Patients with a BMI greater than 40 kg/m2,
7. Patients who abuse of the following substances: alcohol, recreational drugs;
8. Major surgery (e.g. osteotomy) of the index knee within 12 months prior to screening;
9. Minor surgery (e.g. shaving or arthroscopy) of the index knee within 6 months prior to screening;
10. Use of systemic immunosuppressants within 6 weeks prior to screening;
11. Any documented clinically significant degree of cognitive impairment or other condition, finding, or psychiatric illness at screening which, in the opinion of the investigator, could compromise patient safety or interfere with the assessment of the safety and treatment effects of the study injection;

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients with degenerative meniscal tears will be enrolled in the observational study and treated according to the current standard of care which consists in an arthroscopic partial meniscectomy in all the three clinical operative Unit involved in the project.Demographic, anamnestic and clinical data (age, gender, BMI, habits, co-morbidities, pharmacological treatments) of the patients included in the observational clinical study will be collected.
  Clinical routine assessments will be performed before surgery to assess the overall condition of the joint. A morphological profiling based on the MRI will be performed on patients prior or after the surgery since no change in knee morphology is expected to occur. Clinical routine assessments will be performed also after treatment to check for possible joint changes after the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 6-12 months
  To monitor the possible progression of post-meniscectomy OA one year after the treatment
Primary objective | 6-12 months
  Describing the clinical profile of patient
Primary objective | 6-12 months
  Describing the morphological profile of patient
Primary objective | 6-12 months
  Describing the miRNA profile of patient

SECONDARY OUTCOMES:
Secondary objectives | 12 months
  1) To develop the PEARL Patient registry
Secondary objectives | 12 months
  To define specific pre-treatment markers and risk factors related to negative outcome in the long term

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Galeazzi Orthopaedic Institute, Milan, Milano
  - Irccs Humanitas Research Hospital, Milan, Rozzano
  - UNISS Università Degli Studi Di Sassari, Sassari

IPD SHARING:
Plan to Share IPD: Undecided
We are careful not to share patient data from our study and it is necessary that the other centres also agree on approval despite the fact that the Humanitas Research Hospital is the sponsor of the project.

REFERENCES:
- [Background] Allen KD, Thoma LM, Golightly YM. Epidemiology of osteoarthritis. Osteoarthritis Cartilage. 2022 Feb;30(2):184-195. doi: 10.1016/j.joca.2021.04.020. Epub 2021 Sep 14. PMID 34534661
- [Background] Papalia R, Del Buono A, Osti L, Denaro V, Maffulli N. Meniscectomy as a risk factor for knee osteoarthritis: a systematic review. Br Med Bull. 2011;99:89-106. doi: 10.1093/bmb/ldq043. Epub 2011 Jan 19. PMID 21247936

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT06906094/Prot_SAP_000.pdf